CLINICAL TRIAL: NCT06985381
Title: ESAN III - Energy Sensing in Depression Effects of Daucus Carota Subsp. Sativus on Immunomodulation in Patients With Obesity, Depression, and Normal Weight Controls
Brief Title: ESAN III - Energy Sensing in Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ESANIII
Record Dates: First submitted 2025-05-02; First posted 2025-05-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Gut Microbiota Modulation; Immunomodulation
Keywords: Carotenoids; Antioxidant effects; Micronutrient absorption; In-vitro digestion; Intervention study; Nutrition; Natural juice
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The present placebo-controlled, randomized, open, prospective, monocentric study can be classified as a "food product study" (comparison between in trade available carotenoid-rich juice and a placebo).
  Six study groups are designated:
  Group VN = normal weight participants receiving carotenoid-rich juice ("verum") (n=20)
  Group VA = adipose participants receiving carotenoid-rich juice ("verum") (n=20)
  Group VD = depressive patients receiving carotenoid-rich juice ("verum") (n=20)
  Group CN = normal weight participants receiving water (control) (n=20)
  Group CA = adipose participants receiving water (control) (n=20)
  Group CD = depressive patients receiving water (control) (n=20)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Verum Normal Weight Arm (Experimental): Normal weight participants receiving carotenoid-rich juice for 6 weeks.
  Interventions: Other: Carotenoid-rich juice
- Verum Obesity (Experimental): Obese (BMI > 30mg/m2) participants receiving carotenoid-rich juice for 6 weeks
  Interventions: Other: Carotenoid-rich juice
- Control Normal Weight (Placebo Comparator): Normal weight participants receiving control drink (water) for 6 weeks.
  Interventions: Other: Control
- Control Obese (Placebo Comparator): Obese participants receiving control drink (water) for 6 weeks.
  Interventions: Other: Control
- Verum Depression (Experimental): Depressive participants receiving carotenoid-rich natural juice (verum) (n=20).
  Interventions: Other: Carotenoid-rich juice
- Control Depression (Placebo Comparator): Depressive participants receiving water (control) (n=20).
  Interventions: Other: Control

INTERVENTIONS:
Other: Carotenoid-rich juice — The intervention is based on the additional consumption of 200 ml natural carotneoid-rich juice a day for a period of six weeks. The participants are asked to drink the natural and commercially available juice in addition to their regular diet. Further, they are asked not to change their diets and lifestyle behaviour during the intervention.
  Arms: Verum Depression; Verum Normal Weight Arm; Verum Obesity
Other: Control — Participants assigned to the control group are asked to drink additional 200ml of water a day to control liquid intake.
  Arms: Control Depression; Control Normal Weight; Control Obese

SUMMARY:
The purpose of this study is to assess the effects of carotenoids from natural carrot juice on the immune system. Therefore, the study aims to distinguish the effects of natural juices that are rich in phytonutrients such as carotenoids in healthy and depressive individuals, to explore their potential use in therapeutic settings. The consumption of natural fruit juices rich in polyphenols and carotenoids serves as a model for a vegetarian diet, due to the increased micronutrient density derived from plant-based foods. The results obtained may provide preliminary explanatory models for the beneficial effects of a vegetarian diet.

It is hypothesized that the consumption of a natural carotenoid-rich juice alters the expression of regulatory T cells-specific immune cells that contribute to immunomodulation. Furthermore, beneficial changes in the gut microbiome, metabolome, and nutritional status are expected.

This study was registered retrospectively (after recruitment had started) on ClinicalTrials.gov.

ELIGIBILITY:
INCLUSION CRITERIA

Socio-demographic criteria:

* Gender: female
* Age: 18-65 years

Confirmation of study participation:

* Received information on the aims, methods, anticipated benefits, potential risks, and entailed discomforts of the study
* Signed declaration of consent

Subgroup of depressive patients:

* Diagnosis of depression according to the ICD-10 criteria
* Diagnosis confirmed by an experienced psychiatrist

Subgroup of normal weight participants:

• WHO criteria for normal weight (Body Mass Index [BMI] 18.5-24.99 kg/m²)

Subgroup of obese participants:

• WHO criteria for obesity (BMI > 30.0 kg/m²)

EXCLUSION CRITERIA

Formal criteria:

• Lack of informed consent

Health criteria:

* Alcohol or drug abuse
* Acute or chronic diseases or infections (including cancer, fever, pneumological or renal disorders, cardiovascular disease, hematopoietic disorders)
* Digestive disorders (including fructose intolerance, inflammatory bowel disease, irritable bowel syndrome)
* Treatment that may have influenced the microbiome (including antibiotic or antifungal treatment within the previous two months, and daily or irregular intake of prebiotics or probiotics within the previous two months; the intake of yogurt and dairy products is permitted)
* History of gastrointestinal surgery (other than appendectomy)
* Psychiatric disorders (schizophrenia, dementia, bipolar disorder)
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change of baseline regulatory T cells (Tregs) at week 6 (after the intervention) and after a wash-out period at week 12. | From enrollment (baseline) to the end of intervention at week 6 and after a wash-out period at week 12.
  Tregs are involved in modulating the immune system and maintaining tolerance to self-antigens and preventing autoimmune diseases. Regulatory T cells (Treg) will be quantified using multiparameter flow cytometry. Monoclonal antibodies specific for surface markers such as CD3, CD4, CD45RA, CD39 and CD25 will be combined with intracellular anti-Foxp3 for the identification of human Treg.
  Tregs are involved in modulating the immune system and maintaining tolerance to self-antigens and preventing autoimmune diseases. The assessment of Tregs after 12 weeks aims to identify any persisting effects of the intervention.

SECONDARY OUTCOMES:
Effect of carotenoid-rich juice consumption on gut microbiota composition, assessed by changes in alpha diversity (Shannon Index) between intervention and control groups. | From enrollment (baseline) to the end of intervention at week 6 and after a wash-out period at week 12.
Change in plasma carotenoid concentration following carotenoid-rich juice consumption, compared between intervention and control groups. | From enrollment (baseline) to the end of intervention at week 6 and after a wash-out period at week 12.
  Carotenoid plasma concentration is quantified by High-Performance Liquid Chromatography (HPLC).
Change in skin carotenoid levels (measured non-invasively), following carotenoid-rich juice consumption, compared between intervention and control groups. | From enrollment (baseline) to the end of intervention at week 6 and after a wash-out period at week 12.
  Skin carotenoid score is determined on an arbitrary scale non-invasively by spectroscopic devices (Veggimeter and Biozoom). A higher score indicates higher carotenoid content stored in the skin (Score Ranges: Biozoom 0-12M; Veggimeter 0-800).

OTHER OUTCOMES:
Change in depressive symptom severity, as measured by the Beck Depression Inventory-II (BDI-II), from baseline to week 6. | From enrollment (baseline) to the end of intervention at 6 weeks.
  [Range: 0-63; higher scores indicate more severe depressive symptoms.]

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Holasek, Prof, Principal Investigator — Medical University of Graz
Locations (1):
- Medical Universtiy of Graz, Graz, Styria, Austria

REFERENCES:
- [Background] Morkl S, Lackner S, Muller W, Gorkiewicz G, Kashofer K, Oberascher A, Painold A, Holl A, Holzer P, Meinitzer A, Mangge H, Holasek S. Gut microbiota and body composition in anorexia nervosa inpatients in comparison to athletes, overweight, obese, and normal weight controls. Int J Eat Disord. 2017 Dec;50(12):1421-1431. doi: 10.1002/eat.22801. Epub 2017 Nov 13. PMID 29131365
- [Background] Shanahan F, van Sinderen D, O'Toole PW, Stanton C. Feeding the microbiota: transducer of nutrient signals for the host. Gut. 2017 Sep;66(9):1709-1717. doi: 10.1136/gutjnl-2017-313872. Epub 2017 Jun 29. PMID 28663354
- [Background] Kim YS, Sayers TJ, Colburn NH, Milner JA, Young HA. Impact of dietary components on NK and Treg cell function for cancer prevention. Mol Carcinog. 2015 Sep;54(9):669-78. doi: 10.1002/mc.22301. Epub 2015 Apr 1. PMID 25845339
- [Background] Kim W, Lee H. Advances in nutritional research on regulatory T-cells. Nutrients. 2013 Oct 28;5(11):4305-15. doi: 10.3390/nu5114305. PMID 24169507
- [Background] De Rosa V, Galgani M, Santopaolo M, Colamatteo A, Laccetti R, Matarese G. Nutritional control of immunity: Balancing the metabolic requirements with an appropriate immune function. Semin Immunol. 2015 Sep;27(5):300-9. doi: 10.1016/j.smim.2015.10.001. Epub 2015 Oct 29. PMID 26527507